CLINICAL TRIAL: NCT04295070
Title: A Phase 1, First in Human, Randomized, Double-blind, Placebo Controlled Study of the Safety, Tolerability, and Immunogenicity of the CodaVax-RSV Vaccine in Healthy Adult Volunteers
Brief Title: Safety and Immunogenicity of a Live-attenuated Vaccine Against Respiratory Syncytial Virus in Elderly Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Codagenix, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CODA-RSV-001
Record Dates: First submitted 2020-02-28; First posted 2020-03-04 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: RSV; live-attenuated vaccine; codon deoptimized; respiratory infection
MeSH Terms: conditions — Respiratory Syncytial Virus Infections; Respiratory Tract Infections | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Placebo (Placebo Comparator): Saline (0.9%) delivered intranasally via dropper
  Interventions: Biological: Normal saline
- Low dose cohort (Experimental): CodaVax-RSV delivered intranasally via dropper
  Interventions: Biological: CodaVax-RSV
- High dose cohort (Experimental): CodaVax-RSV delivered intranasally via dropper
  Interventions: Biological: CodaVax-RSV

INTERVENTIONS:
Biological: CodaVax-RSV — Codon deoptimized, live-attenuated vaccine against RSV delivered intranasally via dropper
  Arms: High dose cohort; Low dose cohort
Biological: Normal saline — Saline (0.9%) administered via dropper
  Arms: Placebo

SUMMARY:
This Phase I trial will enroll 36 healthy adult volunteers. The study will enroll a sentinel group of 6 younger adults aged 18 to 49 years followed by approximately 30 healthy older adults aged 50 to 75 years. All participants will receive two doses, 28 days apart. The vaccine will be administered as nose drops to both the low and high dose cohorts.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy men and women aged 50 to 75 years of age, inclusive (at the time of informed consent) for the main dosing group or healthy male and female volunteers aged 18 to 49 years of age, inclusive (at the time of informed consent) for the sentinel group;
2. Body mass index (BMI) greater or equal to 18.0 kg/m2 and less than or equal to 35 kg/m2;
3. Participants must be willing to comply with the following conditions to prevent the spread of genetically modified organisms (GMOs) according the Office of the Gene Technology Regulator (OGTR) Licence (DIR 144):

   1. Hygiene measures intended to prevent interpersonal transmission of study drug must be implemented, including but not limited to frequent handwashing with soap or hand disinfectant, respiratory hygiene and cough etiquette within 7 days after each vaccination
   2. Blood, tissue or organs must not be donated within 7 days after each vaccination
   3. Severely immunosuppressed persons who require a protective environment are not to be cared for by the participant within 7 days after each vaccination
   4. Contact is not to be made with severely immunosuppressed persons who require a protective environment within 7 days after each vaccination
   5. All tissues and materials used to collect respiratory secretions for 7 days after each vaccination are to be sealed in a primary container and placed within a secondary container so that it is not accessible to children or animals for 7 days until it is returned to the study site for disposal
4. Adequate venous access for repeated phlebotomies;
5. Screening laboratory results within the normal range or Grade 1 abnormality if the Investigator documents clinical insignificance. Creatine kinase or bilirubin may be Grade 2 if associated with normal alanine aminotransferase (ALT) and aspartate aminotransferase (AST) and the Investigator considers the result not to be clinically significant due to vigorous exercise or Gilbert's syndrome;
6. Negative drug and alcohol screen at Screening (unless explained by prescribed medication);
7. For participants in the main dosing groups, eligible RSV neutralizing antibody titer as defined in the previous seroepidemiology study;
8. Women of childbearing potential (WOCBP) must be non-pregnant and non lactating, and must use an acceptable, highly effective double barrier contraception from Screening until 28 days after the final vaccination. Double contraception is defined as a condom AND one other form of the following:

   * Established hormonal contraception (oral contraceptive pills [OCPs], long acting implantable hormones, injectable hormones);
   * A vaginal ring or an intrauterine device (IUD);
   * Documented evidence of surgical sterilisation at least 6 months prior to screening (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, or bilateral oophorectomy for women or vasectomy for men [with appropriate post vasectomy documentation of the absence of sperm in semen] provided the male partner is a sole partner) Women not of childbearing potential must be postmenopausal for greater or equal to 12 months. Postmenopausal status will be confirmed through testing of follicle stimulating hormone (FSH) levels greater or equal to 40 IU/mL at Screening for amenorrhoeic female participants.

   Females who are abstinent from heterosexual intercourse will also be eligible. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post ovulation methods) and withdrawal are not considered highly effective methods of birth control.

   Female participants who are in same sex relationships are not required to use contraception.

   WOCBP must have a negative pregnancy test at Screening and Day 1 and be willing to have additional pregnancy tests as required throughout the study;

   Males must be surgically sterile (>30 days since vasectomy with no viable sperm), abstinent, or if engaged in sexual relations with a WOCBP, his partner must be surgically sterile (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy, bilateral oophorectomy) or using an acceptable, highly effective double barrier contraceptive method from Screening until until 28 days after the final vaccination. Acceptable methods of double barrier contraception include the use of condoms AND the use of an effective contraceptive for the female partner that includes: OCPs, long-acting implantable hormones, injectable hormones, a vaginal ring or an IUD. Participants with same sex partners (abstinence from penile-vaginal intercourse) are eligible when this is their preferred and usual lifestyle.
9. Males must not donate sperm for at least 90 days after the final vaccination;
10. Participants must have the ability and willingness to attend the necessary visits to the clinical research unit (CRU);
11. Participants must be willing and able to provide written informed consent prior to the commencement of any study procedures.

Exclusion Criteria:

1. Pregnant or lactating at Screening or planning to become pregnant (self or partner) prior to 28 days after the final vaccination;
2. Household contacts or caregivers of infants < 12 months of age or immunocompromised individuals (for the period up through 28 days post final vaccination). Immunocompromised individuals defined as but not limited to:

   1. Persons who are human immunodeficiency virus (HIV)-infected
   2. Persons who have received chemotherapy within 6 months
   3. Persons receiving immunosuppressive agents
   4. Person living with solid organ or bone marrow transplant;
3. Positive result for HIV, hepatitis B virus (HBV), or hepatitis C virus (HCV) at Screening;
4. Asthma or other chronic lung disease that is greater than mild in severity. Specifically excluded are participants with any of the following history related to asthma or lung disease:

   1. Daily symptoms for more than 1 week in the past 5 years;
   2. Use of short acting beta 2 agonists in the past 5 years (e.g., albuterol);
   3. Use of inhaled steroids, theophylline or pulse systemic steroids in the past 5 years; or
   4. Any history of intubation or hospitalization related to asthma or other chronic lung disease.
5. History of diabetes mellitus (gestational diabetes is allowed if treatment was not required postpartum and serum glucose is currently within the normal range);
6. History of coronary artery disease, arrhythmia, or congestive heart failure;
7. Clinically significant ECG abnormality as determined by the Investigator at Screening;
8. Poorly controlled hypertension (systolic blood pressure >150 mmHg or diastolic blood pressure >95 mmHg) at Screening or predose on Day 1;
9. History of anaphylaxis or angioedema;
10. History of severe reaction to immunization;
11. Known allergy to any of the ingredients in the vaccine formulation;
12. History of chronic rhinitis, nasal septal defect, cleft palate, nasal polyps, or other nasal abnormality that might alter nasal mucosa and affect vaccine response;
13. Previous nasal surgery or nasal cauterization;
14. Epistaxis (nosebleed), symptoms of upper respiratory infection or subjective fever or malaise within 3 days prior to dosing on Day 1 (temporary exclusion criterion);
15. Any symptoms or signs on Day 1 that could inhibit the proper administration of the investigational product (IP) or interpretation of solicited AEs diary (e.g., temperature >38°C, nasal congestion or rhinorrhea) (temporary exclusion criteria);
16. Known or suspected malignancy, except for non-melanoma skin cancers and other early stage surgically excised malignancies that the Investigator considers to be exceedingly unlikely to recur;
17. Immunodeficiency including the use of corticosteroids (including IN steroids), alkylating drugs, antimetabolites, radiation, immune-modulating biologics, or other immunomodulating therapies within 90 days prior to dosing on Day 1, or for those participants that plan to use any of these during the study follow-up period. Topical steroid creams used on the skin are allowed;
18. History of bleeding disorder (e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions);
19. History of autoimmune or demyelinating illness;
20. History of psychosis, hospitalization for psychiatric illness, or suicide attempt in the past 10 years;
21. History of seizures (other than childhood febrile seizures), dementia or progressive neurological disease;
22. Receipt of IN medications (including over the counter [OTC] medications but excluding saline) within 30 days prior to Day 1;
23. Receipt of any other IP within 30 days or 5 half lives (whichever is longer) prior to Day 1;
24. Receipt of any vaccine, tuberculosis (TB) skin test or allergy antigen inoculations within 30 days prior to Day 1 or planned up to Day 57;
25. Receipt of IN vaccine within 90 days prior to Day 1;
26. Receipt of any licensed or investigational RSV vaccine;
27. Receipt of blood transfusion or blood products within 90 days prior to Day 1 or planned up through Day 57;
28. Planned elective hospitalization or surgical procedure through Day 57;
29. Other chronic medical conditions not mentioned must be stable without necessitating medication changes within 30 days prior to Day 1;
30. Past regular use or current use of IN illicit drugs;
31. Smokers of any type (e.g., cigarettes, electronic cigarettes, marijuana). Prior smokers must have quit smoking at least 30 days prior to Day 1;
32. Employee of Codagenix, vendors, or research sites associated with the study;
33. Any medical, psychiatric or social condition, or occupational or other responsibility that, in the judgment of the Investigator, would interfere with or serve as a contraindication to protocol adherence, assessment of safety (including reactogenicity), or a participant's ability to give informed consent.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-07-10 (Actual); Primary Completion 2021-03-06 (Actual); Study Completion 2021-05-26 (Actual)

PRIMARY OUTCOMES:
Reactogenicity counts | Days 1 through 7
  Counts of participants with local and systemic events along with symptom severity and duration
Reactogenicity percentages | Days 1 through 7
  Percentages of participants with local and systemic events along with symptom severity and duration
Adverse events counts | Days 1 through 57
  Counts of participants with AEs not included as reactogenicity events
Adverse events percentages | Days 1 through 57
  Percentages of participants with AEs not included as reactogenicity events
Serious adverse events | Days 1 through 209
  Number of medically-attended AEs (MAEs), new onset chronic illnesses (NCIs), and serious AEs (SAEs) will be captured

SECONDARY OUTCOMES:
RSV-specific IgG | Days 1, 15, 29, 43, 57, 113, and 209
  Titer of RSV-specific immunoglobulin G (IgG) antibodies measured by enzyme-linked immunosorbent assay (ELISA) in serum
Seroconversion rate IgG | Days 1, 15, 29, 43, 57, 113, and 209
  Percent of participants with at least 4-fold increase in RSV-specific IgG as measured by ELISA over baseline
Neutralizing antibodies | Days 1, 15, 29, 43, 57, 113, and 209
  Titer of neutralizing antibodies in serum measured via RSV micro neutralization assay
Percent of patients seroconverting via neutralizing antibodies | Days 1, 15, 29, 43, 57, 113, and 209
  Percent of participants with at least 4- fold increase in neutralizing antibodies in serum over baseline
RSV-specific IgA | Days 1, 15, 29, 43 and 57
  Geometric mean titer (GMT) of antibodies measured by ELISA in nasopharyngeal (NP) swab specimens
Percent of patients seroconverting via IgA | Days 1, 15, 29, 43 and 57
  Percent of participants with at least 4 fold increases in RSV-specific IgA over baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Nucleus Network/Q-Pharm, Brisbane, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No